CLINICAL TRIAL: NCT02578537
Title: COmparison of the Pharmacodynamics and Pharmacokinetics of Ticagrelor Versus Clopidogrel in Patients With Chronic Kidney Disease and Non-ST-Elevation Acute Coronary Syndromes(OPT-CKD Trial)
Brief Title: COmparison of the Pharmacodynamics and Pharmacokinetics Ticagrelor Versus Clopidogrel in Patients With CKD and NSTE-ACS
Acronym: OPT-CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Dr, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-14-10607
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome; Chronic Kidney Disease
Keywords: Ticagrelor; Pharmacokinetics; NSTE-ACS; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor group (Experimental): ticagrelor 180mg loading, followed by 90mg bid for 30 days
  Interventions: Drug: Ticagrelor
- Clopidogrel group (Active Comparator): clopidogrel 600mg loading, followed by 75mg/d for 30 days
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor group:all patients receive ticagrelor (180 mg loading dose, then 90 mg twice daily followed for 30 days). All patients were given aspirin 100 mg per day unless they were intolerant. For those not previously given aspirin, a loading dose of 300 mg was preferred.
  Other Names: Brilinta
  Arms: Ticagrelor group
Drug: Clopidogrel — Clopidogrel group:all patients receive clopidogrel (600 mg loading dose, then 75 mg once daily followed for 30 days). All patients were given aspirin 100 mg per day unless they were intolerant. For those not previously given aspirin, a loading dose of 300 mg was preferred.
  Other Names: Plavix
  Arms: Clopidogrel group

SUMMARY:
Ticagrelor, a new P2Y12 receptor antagonist, achieve faster, consistent and higher platelet inhibition than clopidogrel, which was considered more noticeable in patients with ACS combining chronic kidney disease(CKD). Nonetheless, the pharmacokinetic properties of ticagrelor in the patients with CKD and NSTE-ACS has not been thoroughly studied. This study was designed to provide PK and PD data of ticagrelor compared with clopidogrel, in order to estimate that ticagrelor is superior to clopidogrel in getting better inhibition of platelet in patients with CKD and NSTE-ACS. P2Y12 inhibitor naïve patients with CKD (eGFR < 60 ml/min/1.73m2 ) and NSTE-ACS will be enrolled in this single-center, prospective, randomized, parallel-control study and randomly assigned in a one-to-one ratio to receive ticagrelor or clopidogrel on top of chronic aspirin treatment. The primary endpoint was the PRU by Verify Now at 30 days after loading dose.

DETAILED DESCRIPTION:
Dual antiplatelet therapy with aspirin and clopidogrel has become the standard care in patients with acute coronary syndrome (ACS). However, clopidogrel is being questioned for its insufficient platelet inhibition and residual platelet reactivity, especially in patients with impaired renal function. Ticagrelor, a new P2Y12 receptor antagonist, achieve faster, consistent and higher platelet inhibition than clopidogrel, which was more noticeable in patients with ACS combining chronic kidney disease(CKD). Nonetheless, the pharmacokinetic properties of ticagrelor in the patients with CKD and NSTE-ACS, to the best of the investigators' knowledge, has not been thoroughly studied. This study was designed to provide PK and PD data of ticagrelor compared with clopidogrel, in order to estimate that ticagrelor is superior to clopidogrel in getting better inhibition of platelet in patients with CKD and NSTE-ACS. The potential hypothesis is to evaluate the correlation of platelet inhibition and renal function and CYP2C19 gene type in patients treated by ticagrelor and clopidogrel. P2Y12 inhibitor naïve patients with CKD (eGFR < 60 ml/min/1.73m2 ) and NSTE-ACS will be enrolled in this single-center, prospective, randomized, parallel study and randomly assigned in a one-to-one ratio to receive ticagrelor or clopidogrel on top of chronic aspirin treatment. The primary endpoint was the PRU by Verify Now at 30 days after loading dose.

ELIGIBILITY:
Inclusion Criteria:

* P2Y12 inhibitor naïve patients presenting with NSTE-ACS (unstable angina or non-ST segment elevation myocardial infarction).
* Males and non-pregnant females > 18 years of age.
* eGFR<60 ml/min/1.73m2 (MRDR formula).
* With planned percutaneous coronary intervention(PCI will be performed over 24 hours after loading dose).
* Written informed consent provided.Provision of informed consent prior to any study specific procedures.

Exclusion Criteria:

* Cardiogenic shock.
* Thrombolytic therapy administered before randomization.
* Active bleeding or bleeding predisposition, including the retinal or vitreous hemorrhage , gastrointestinal or urinary tract hemorrhage , history of intracranial haemorrhage or cerebral infarction .
* Hypersensitivity to ticagrelor or any excipients.
* Deep puncture or major surgery within 1 month.
* Untreated or uncontrolled hypertension with blood pressure >180/110 mmHg.
* Known hemoglobin <10 g/dL or platelet count <100 × 109/L.
* Known moderate or severe hepatic impairment.
* Known aminotransferase level >3x the upper limit of normal.
* Known allergy to any of the study drugs or devices (aspirin, clopidogrel, ticagrelor stainless steel, contrast agents, etc.).
* Pregnancy or lactation.
* Any condition which might interfere with study compliance, or otherwise unsuitable for study participation as judged by the investigators.
* Unwilling or unable to get repeat platelet assay or clinical follow-up.
* Unwilling or unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
PRU assayed by VerifyNow | 30 days after loading does of study drug

SECONDARY OUTCOMES:
PRU assayed by VerifyNow | at the time of pre-dose, and 2 hours, 8 hours, and 24 hours after loading dose of study durg.
Index of Platelet activity | at the time of 2 hours, 8 hours, and 24 hours after loading dose of study drug
  calculated by the change of the P2Y12 reaction units (PRU) from baseline
Rate of high on-treatment platelet reactivity (HPR) | at the time of pre-dose, and 2 hours, 8 hours, 24 hours and 30 days after loading dose of study durg.
Plasma concentration of ticagrelor and clopidogrel | at 2 hours, 8 hours, and 24 hours after loading dose of study durg.
Bleeding events | 30 days after loading does of study drug
  by BARC classification

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730